CLINICAL TRIAL: NCT03914391
Title: To Identify Potential New Urine Markers for the Screening of Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, NG Chi Fai, Professor, Chinese University of Hong Kong
Other Study IDs: CRE-2018.376
Record Dates: First submitted 2019-04-09; First posted 2019-04-16 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prostate gland is a clinically important male sexual organ and its main function is for the production of semen. Globally, it is the second most common cancer in men globally and is also the fifth cancer cause for death in male. Despite the improvement in the understanding of prostate cancer, the current usage of serum prostate specific antigen (PSA) as a diagnostic marker is still not ideal. Many patients with elevated PSA and then subjected to prostate biopsy were found to have no prostate cancer. Therefore, there is a need to discover new biological markers to improve the current situation in diagnosis and also management of prostate cancer.

From the earlier small-scale studies, urinary spermine levels have been shown to correlate well with prostate cancer diagnosis and cancer aggressiveness. Due to its nature, it could provide a more convenient and non-invasive method for detecting prostate cancer. The purpose of this study was to collect urine samples to study the role of potential new urine diagnostic markers (including Spermine and others) for prostate cancer diagnosis.

DETAILED DESCRIPTION:
Prostate cancer (PC) is highly prevalent worldwide and is the second most commonly diagnosed cancer in men globally and is the 5th leading cause of cancer death in men. 1 In some Asian areas, even n with widely used serum Prostate Specific Antigen (PSA) diagnostic testing, more than 50% men with newly diagnosed PC are deemed to have high risk disease. 2 However, the current use of serum PSA as a diagnostic marker is unsatisfactory. Many patients has elevated serum PSA is actually due to other causes and also the level of serum PSA do not correlate with the staging and grading of prostate cancer. 3 Moreover, the use of serum PSA required blood taking which is invasive and non-convenience for large scale screening. Therefore, newer markers is needed for more simple and accurate diagnosis of prostate cancer.

One example of such cancer biomarkers are natural polyamines. Interests on these analytes have been starting in 1971 when Russell reported a considerable increase of urinary polyamines such as putrescine (Put), spermidine (Spd) and spermine (Spm) in patients with various types of solid tumors and leukaemias. 4 Afterwards, polyamine studies focusing on specific cancers continued, like cervical cancer, 5 colorectal cancer 6 and breast cancer, 7 etc. In investigators' recent study, investigators have explored the potential roles of urinary polyamines as prostate cancer biomarkers were evaluated. Patients with prostate cancer (PCa), benign prostatic hyperplasia (BPH) patients and healthy controls (HC) showing PSA>4.0ng/ml were enrolled in the study.8 Their urine samples were obtained, and the urinary levels of Put, Spd, Spm were determined by ultra-high-performance liquid chromatography coupled with triple quadrupole mass spectrometer (UPLC-MS/MS). Receiver operating characteristics (ROC) curve and Student's t- test were used to evaluate their diagnostic accuracies. Among the three biogenic polyamines, Spm had demonstrated a good diagnostic performance when comparing their levels in PCa patients with BPH patients (1.47 in PCa vs 5.87 in BPH; p<0.0001). The results were in accordance with transrectal ultrasound prostatic biopsy (TRUSPB) results, with an area under curve (AUC) value of 0.83±0.03. Therefore, urinary Spm could have a potential to serve as a novel PCa diagnostic biomarker, which in turn could help to address the limited sensitivity and specificity problem of serum PSA test.

Therefore, investigators would like to have a larger scale study, with inclusion of subjects from different geographic locations, to further assess the correlation spermine and other potential newer urine markers with diagnosis of prostate cancer and investigate their role as a potential non-invasive marker for prostate cancer risk stratification and prognosis prediction.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male patients with age > 18 years old
2. Subject has elevated serum PSA level above 4ng/ml
3. Clinical planned for prostatic biopsy.

Exclusion Criteria:

1. Patient with recent urinary tract infection within 6 weeks prior to PSA testing and urine collection.
2. Patient with recent urethral instrumentation, such as Foley catheter insertion, cystoscopy etc, within 6 weeks prior to PSA testing and urine collection.
3. Patient with consumption of 5 alpha reductase inhibitors in past 6 months.
4. Patient did not receive any surgery for prostatic pathology
5. Patient refused or unable to provide consent for the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients who has elevated serum PSA, i.e. > 4ng/ml, and planned for prostatic biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To investigate the role of urine spermine in the diagnosis of prostate cancer | Baseline (one-time point)
  Fresh urine will be collected for liquid chromatography and mass spectrometry to detect the concentration of spermine in urine. Then the The correlation between the concentration of urine spermine and serum PSA level and pathological result will be assessed.
To investigate the role of urine spermine in prognostic prediction of prostate cancer | Baseline (one-time point)
  Fresh urine will be collected for liquid chromatography and mass spectrometry to detect the concentration of spermine in urine. Then the The correlation between the concentration of urine spermine and pathological result and serum PSA level will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai Ng, MD, Principal Investigator — The Chinese University if Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong